CLINICAL TRIAL: NCT04258345
Title: Artificially Sweetened Beverage Feeding Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not yet funded
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Yasmin Mossavar-Rahmani, Principal Investigator, Albert Einstein College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-11111
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Feeding Arm (Other): This is a feeding study.
  Interventions: Other: ASB Feeding Study

INTERVENTIONS:
Other: ASB Feeding Study — Participants will undergo a washout period and then scheduled for blood draw after which ASB feeding period will begin followed by a second blood draw.

SUMMARY:
The aims of the study are to conduct a pre- and post- two week feeding study of artificial sweetened beverage consumption in middle-aged women. The study will also compare metabolic profiles before and after artificially sweetened beverage consumption.

DETAILED DESCRIPTION:
The aims of the study are to:

1. To conduct a pre- and post- two week feeding study of Artificially Sweetened Beverage (ASB) in women.
2. To assess the general levels of ASB consumption.
3. To compare metabolic profiles before and after beverage consumption

ELIGIBILITY:
Inclusion Criteria:

• Healthy women

Exclusion Criteria:

• Having a history of diabetes or cardiovascular disease and any other health or chronic condition that precludes participation in the study.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 0 (Actual)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Change in artificial sweetener levels pre- and post- feeding | two weeks
  Change in metabolites pre- and post-feeding

IPD SHARING:
Plan to Share IPD: No
Not at this time.